CLINICAL TRIAL: NCT01121627
Title: Effects of Computer-based Cognitive Training on Gait Function in Individuals With Parkinson Disease
Brief Title: Computer-based Cognitive Training for Parkinson Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clalit Health Services (Other)
Collaborators: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, Uzi Milman, Director, Clinical Research Unit, Clalit Health Services, Haifa and Western Galilee District and the Department of Family Medicine, Faculty of Medicine, Technion- Israel Institute of Technology, HAIFA, ISRAEL., Clalit Health Services
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K-10-0036-ctil
Record Dates: First submitted 2010-05-10; First posted 2010-05-12 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Parkinson Disease; Gait
Keywords: Computerized Cognitive training; Quality of life; Gait Function; Executive Function
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Computerized cognitive training (Experimental): A 12 week computerized cognitive training
  Interventions: Other: Computerized cognitive training

INTERVENTIONS:
Other: Computerized cognitive training — A 12 week computerized cognitive training at home with the Attengo™ software program.

SUMMARY:
Parkinson's Disease (PD) is a neurodegenerative, progressive illness. It is a multi-system disease that influences not only the motor but also the cognitive and autonomic systems. The main cognitive impairment in individuals with PD is found in executive function (EF). EF is defined as a set of cognitive skills necessary for planning, monitoring and executing sequences of complex activities.

The primary study hypothesis is that computer-based training aimed at improving executive function will have a beneficial effect on gait functions.

DETAILED DESCRIPTION:
Parkinson Disease (PD) is a neurodegenerative, progressive illness. It is a multi-system disease that influences not only the motor but also the cognitive and autonomic systems. The main cognitive impairment in individuals with PD is found in executive function (EF). EF is defined as a set of cognitive skills necessary for planning, monitoring and executing sequences of complex activities. Previous studies have revealed some relation between cognitive states and physical functions in healthy adults. Few studies have examined the effect of computer-based cognitive training on various populations. These studies showed a positive emotional-cognitive effect in those populations. This type of intervention plan was also applied to PD patients. However, there are no reports on the effect of intentional cognitive training on gait functions. The purpose of the study is to assess whether cognitive training, designed to improve EF ability, can also improve gait function in PD patients.

ELIGIBILITY:
Inclusion Criteria:

1. Idiopathic PD.
2. Aged 50-80, living in north region of Israel.
3. Receive regular medications for PD.
4. Not suffering from irregular cognitive disturbance or MMSE<25.
5. Measured 1-3 on the Hoehn & Yahr scale.
6. Have access to a computer and the ability to operate it.

Exclusion Criteria:

1. Brain operation, including DBS transplant.
2. History of orthopedic problems that can impair gait (hip/knee fractures and back problems).
3. Orthopedic operation on lower limbs performed no later than six months prior to the beginning of the study.
4. Unbalanced general health: uncontrolled diabetes or blood pressure, etc.
5. Inability to walk independently.
6. Immunodeficiency diseases, active cancer, ischemic diseases.
7. Vision impairment, partial/full blindness.
8. Having participated in similar research or cognitive assessment during the previous year.
9. Have received cognitive or gait training under physical therapy or other programs.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-07; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Gait Function | 18 weeks
  At enrollment eligible individuals will undergo a thorough baseline assessment using a predefined set of tests and performance measurements. Within a week after enrollment each individual will receive guided training on the use of the intervention tool, the Attengo™ software program. Thereafter they will train at their homes, at least three times a week, for a period of 12 weeks. Follow up assessments will be performed within a week of the end of the training period and 4 weeks thereafter to check for long-term cognitive and motor changes.

SECONDARY OUTCOMES:
Executive function | 18 weeks
  At enrollment eligible individuals will undergo a thorough baseline assessment using a predefined set of tests and performance measurements. Within a week after enrollment each individual will receive guided training on the use of the intervention tool, the Attengo™ software program. Thereafter they will train at their homes, at least three times a week, for a period of 12 weeks. Follow up assessments will be performed within a week of the end of the training period and 4 weeks thereafter to check for long-term cognitive and motor changes.
Quality of life. | 18 weeks
  At enrollment eligible individuals will undergo a thorough baseline assessment using a predefined set of tests and performance measurements. Within a week after enrollment each individual will receive guided training on the use of the intervention tool, the Attengo™ software program. Thereafter they will train at their homes, at least three times a week, for a period of 12 weeks. Follow up assessments will be performed within a week of the end of the training period and 4 weeks thereafter to check for long-run cognitive and motor changes.

CONTACTS AND LOCATIONS:
Overall Officials: Uzi Milman, MD, Principal Investigator — Clalit Health Services; Jeffrey M Hausdorff, PhD, Principal Investigator — Tel-Aviv Sourasky Medical Center; Anat Mirelman, Phd, Principal Investigator — Tel-Aviv Sourasky Medical Center; Hagit Atias, BA, Principal Investigator — Clalit Health Services
Locations (1):
- Clalit Health Services, Haifa and Western Galilee District, Haifa, Israel

REFERENCES:
- [Result] Milman U, Atias H, Weiss A, Mirelman A, Hausdorff JM. Can cognitive remediation improve mobility in patients with Parkinson's disease? Findings from a 12 week pilot study. J Parkinsons Dis. 2014;4(1):37-44. doi: 10.3233/JPD-130321. PMID 24322063